CLINICAL TRIAL: NCT05086900
Title: Developing a Patient Reported Outcome Measure for Recurrent Urinary Tract Infection
Brief Title: Developing a PROM for Recurrent Urinary Tract Infection
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Reading (Other)
Collaborators: Live UTI Free (Unknown); University of Buckingham (Unknown)
Responsible Party: Principal Investigator, Katherine Finlay, Lecturer in Psychology, University of Reading
Other Study IDs: RUTI01-KF-2021
Record Dates: First submitted 2021-08-17; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Urologic Diseases; Patient Satisfaction; Pain, Chronic; Sexual Dysfunction
Keywords: urinary; UTI; burden; outcome measure
MeSH Terms: conditions — Urologic Diseases; Patient Satisfaction; Chronic Pain; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional Cross-sectional Patient Reported Outcome Measure Development — Development of Patient Reported Outcome Measure

SUMMARY:
This study aims to develop and validate the first set of patient-reported outcome measures for recurrent urinary tract infection (UTI): the Recurrent UTI Symptom Scale and the Recurrent UTI Impact Questionnaire. These tools could be used in clinical practice, clinical trials and research to gather an insight into a patient's perspective of their recurrent UTI symptom severity and its impact on their life, as well as determining any possible improvement or other change in their condition due to interventions (e.g. antibiotic treatment).

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is a highly prevalent infection, most frequently affecting females. Recurrent UTI, a chronic condition defined as experiencing two or more UTIs in six months or three or more in twelve months, is associated with significant symptom burden and lowered quality of life. In addition to this personal impact, the effects span more widely to issues such as increased healthcare costs, work absenteeism, and antimicrobial resistance.

There are currently no validated patient-reported outcome measures to assess recurrent UTI symptoms and impact. These measures are much needed to encourage a more patient-centred approach to recurrent UTI treatment and care, which could be especially important given evidence that current routine testing approaches, and thus treatment approaches, are not sufficient alone.

This mixed-methods study aims to consult both clinicians and patients in order to develop and validate the first set of patient-reported outcome measures for recurrent UTI.

Outline:

Phase I: Concept elicitation Conduct a literature review and examine the findings of an international qualitative study exploring the experience of over 2,000 people living with recurrent UTI.

Phase II: Initial development and item generation Develop draft questionnaire items, instructions, and scale response options in line with current healthcare guidance and conclusions from Phase I.

Phase III: Modified Delphi method with 10-20 expert clinicians Screen the draft questionnaires by two rounds of a modified Delphi method, assessing item and instruction clarity and relevance for recurrent UTI.

Use qualitative comments, content validity indices, and consensus scores to refine existing items, and remove or add new ones where appropriate.

Phase IV: Cognitive interviews with 25-30 patients Conduct one-to-one cognitive interviews using a think aloud and verbal probing procedure to verify the content validity and clarity of the new measures from the patient's perspective.

Summarise and analyse the interview transcripts using the Questionnaire Appraisal System and content analysis, used to refine the measures before Phase V.

Phase V: Two-part online pilot with 100+ patients Conduct a cross-sectional survey in which participants complete the new recurrent UTI measures and comparable existing standardised measures for each subscale (e.g. UTI Symptom Assessment). Participants will complete this twice, 24 hours apart.

Verify the psychometric properties of the new measures, including exploratory factor analysis, internal consistency, test-retest reliability, and criterion validity.

Optimise the measures for clinical and research purposes based on these analyses.

ELIGIBILITY:
Inclusion Criteria:

Clinicians:

* Aged at least 18 years old.
* Specialist doctor or nurse in the field of urology or a closely related discipline OR general health doctor or nurse.
* Minimum of 3 years of direct experience treating patients with recurrent UTI.

Patients:

* Aged at least 18 years old.
* Experiences recurrent UTI as defined by the European Association of Urology: minimum of 2 UTIs in 6 months or minimum of 3 UTIs in 12 months.

Exclusion Criteria:

Patients:

* Current diagnosis of interstitial cystitis.
* Non-fluent or non-advanced level of English.
* Current pregnancy.
* Current use of urinary catheterisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the target patient population consists of adults with a minimum of 2 UTIs in 6 months or a minimum of 3 UTIs in 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Recurrent Urinary Tract Infection Symptom Scale | Baseline (Time 1)
  RUTISS; Total minimum score = 0, total maximum score = 170. Newly designed instrument that can measure the patient experience of recurrent UTI symptoms and pain and/or discomfort; Urinary symptoms sub-scale minimum score = 0, maximum score = 70; urinary pain sub-scale minimum score = 0, maximum score = 100; higher scores indicate higher symptom severity
Recurrent Urinary Tract Infection Symptom Scale | Time 2 (24 hours after baseline)
  RUTISS; Total minimum score = 0, total maximum score = 170. Newly designed instrument that can measure the patient experience of recurrent UTI symptoms and pain and/or discomfort; Urinary symptoms sub-scale minimum score = 0, maximum score = 70; urinary pain sub-scale minimum score = 0, maximum score = 100; higher scores indicate higher symptom severity
Recurrent Urinary Tract Infection Impact Questionnaire | Baseline (Time 1)
  RUTIIQ; Total minimum score = 0, maximum score = 300. Higher scores indicate higher rUTI impact and psychosocial burden. Newly designed instrument that can measure the patient experience of recurrent UTI impact on personal wellbeing, social activities, work and daily activities, sexual activity, and satisfaction with UTI-related medical care; personal wellbeing sub-scale minimum score = 0; maximum score = 40; social wellbeing sub-scale minimum score = 0, maximum score = 40; work/activity interference sub-scale minimum score = 0, maximum score = 70; sexual wellbeing sub-scale minimum score = 0, maximum score = 40; patient satisfaction sub-scale minimum score = 0, maximum score = 100.
Recurrent Urinary Tract Infection Impact Questionnaire | Time 2 (24 hours after baseline)
  RUTIIQ; Total minimum score = 0, maximum score = 300. Higher scores indicate higher rUTI impact and psychosocial burden. Newly designed instrument that can measure the patient experience of recurrent UTI impact on personal wellbeing, social activities, work and daily activities, sexual activity, and satisfaction with UTI-related medical care; personal wellbeing sub-scale minimum score = 0; maximum score = 40; social wellbeing sub-scale minimum score = 0, maximum score = 40; work/activity interference sub-scale minimum score = 0, maximum score = 70; sexual wellbeing sub-scale minimum score = 0, maximum score = 40; patient satisfaction sub-scale minimum score = 0, maximum score = 100.

SECONDARY OUTCOMES:
Urinary Tract Infection Symptom Assessment | Baseline (Time 1)
  (UTISA) 7 items assessing the severity of UTI symptoms in the past 24 hours; minimum total score = 0; maximum total score = 21. Higher scores indicate higher symptom severity and clinical cut-off for presence of a UTI = 3.
Urinary Tract Infection Symptom Assessment | Time 2 (24 hours after baseline)
  (UTISA) 7 items assessing the severity of UTI symptoms in the past 24 hours; minimum total score = 0; maximum total score = 21. Higher scores indicate higher symptom severity and clinical cut-off for presence of a UTI = 3.
Numerical Pain Rating Scale | Baseline (Time 1)
  Minimum total score = 0, maximum total score = 10. Higher scores indicate higher pain intensity. Scores assess pain intensity in the past 24 hours
Numerical Pain Rating Scale | Time 2 (24 hours after baseline)
  Minimum total score = 0, maximum total score = 10. Higher scores indicate higher pain intensity. Scores assess pain intensity in the past 24 hours
Depression | Baseline (Time 1)
  Patient Health Questionnaire-9; Minimum total score = 0, maximum total score = 27; higher scores indicate higher depression levels.
Depression | Time 2 (24 hours after baseline)
  Patient Health Questionnaire-9; Minimum total score = 0, maximum total score = 27; higher scores indicate higher depression levels.
Anxiety | Baseline (Time 1)
  Generalised Anxiety Disorder - 7; minimum total score = 0, maximum total score = 21. Higher scores indicate higher anxiety severity.
Anxiety | Time 2 (24 hours after baseline)
  Generalised Anxiety Disorder - 7; minimum total score = 0, maximum total score = 21. Higher scores indicate higher anxiety severity.
Loneliness | Baseline (Time 1)
  UCLA Loneliness Scale (V3); minimum total score = 0, maximum total score = 80; Higher scores indicate greater feelings of loneliness/social isolation.
Loneliness | Time 2 (24 hours after baseline)
  UCLA Loneliness Scale (V3); minimum total score = 0, maximum total score = 80; Higher scores indicate greater feelings of loneliness/social isolation.
Work Productivity and Impairment Questionnaire | Baseline (Time 1)
  Measure assessing specific health problems impairing work capacity. Work impairment sub-scale minimum score = 0; maximum work impairment = 100; activity impairment minimum total score = 0, maximum activity impairment = 100. Higher scores indicate greater impairment due to health problems.
Work Productivity and Impairment Questionnaire | Time 2 (24 hours after baseline)
  Measure assessing specific health problems impairing work capacity. Work impairment sub-scale minimum score = 0; maximum work impairment = 100; activity impairment minimum total score = 0, maximum activity impairment = 100. Higher scores indicate greater impairment due to health problems.
Sexual Distress | Baseline (Time 1)
  Female Sexual Distress Scale for assessing feelings of sexual distress. Minimum total score = 0, maximum total score = 52. Higher scores indicate greater sexual distress. Scores greater than 10 may indicate atypical/abnormal sexual distress.
Sexual Distress | Time 2 (24 hours after baseline)
  Female Sexual Distress Scale for assessing feelings of sexual distress. Minimum total score = 0, maximum total score = 52. Higher scores indicate greater sexual distress. Scores greater than 10 may indicate atypical/abnormal sexual distress.
Satisfaction with Treatment | Baseline (Time 1)
  Patient Satisfaction Questionnaire - 18: 18 items assessing feelings about current medical care. Higher scores indicate greater satisfaction with medical care. Minimum total score = 18; maximum total score = 90.
Satisfaction with Treatment | Time 2 (24 hours after baseline)
  Patient Satisfaction Questionnaire - 18: 18 items assessing feelings about current medical care. Higher scores indicate greater satisfaction with medical care. Minimum total score = 18; maximum total score = 90.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Finlay, PhD, Study Director — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Newlands AF, Roberts L, Maxwell K, Kramer M, Price JL, Finlay KA. Development and psychometric validation of a patient-reported outcome measure of recurrent urinary tract infection impact: the Recurrent UTI Impact Questionnaire. Qual Life Res. 2023 Jun;32(6):1745-1758. doi: 10.1007/s11136-023-03348-7. Epub 2023 Feb 6. PMID 36740638

DOCUMENTS (1):
  • Informed Consent Form (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT05086900/ICF_000.pdf